CLINICAL TRIAL: NCT06280482
Title: Nicotinamide Riboside (NR) to Treat Moyamoya-like Cerebrovascular Disease in Smooth Muscle Dysfunction Syndrome (SMDS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Dianna M Milewicz, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0332
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Smooth Muscle Dysfunction Syndrome (SMDS)
Keywords: smooth muscle aortic alpha-actin (ACTA2); arginine 179 residue; Nicotinamide Riboside; Stroke; Cerebrovascular Disease; Thoracic Aortic Aneurysms and Dissections
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Aortic Aneurysm, Thoracic | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Nicotinamide riboside (NR)

INTERVENTIONS:
Drug: Nicotinamide riboside (NR) — Participants will take their weight-based dose of NR once daily by mouth with food for 60 days.

SUMMARY:
The purpose of this study is to determine whether SMDS patients treated with NR at the proposed dose exhibit decreased glucose uptake in the aorta, to determine if NR treatment results in measurable changes of blood NAD+ and NR levels, to determine if aortic measurements are stable after treatment with NR and to evaluate the safety and tolerability of NR in SMDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with SMDS with confirmed ACTA2 mutation disrupting arginine 179
* Parental/guardian permission (informed consent) and, if appropriate, child assent.

Exclusion Criteria:

* Individuals who have undergone surgery to replace aneurysmal or dissected ascending and root aortic tissue with a graft.
* Additional medical conditions that impair the patient's ability to participate in the study.
* Known allergy or sensitivity to niacin or nicotinamide riboside.
* Prior consumption of niacin or nicotinamide riboside supplement within the prior eight weeks.
* Failure to provide informed consent.
* Concurrent participation in another intervention trial.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood | Baseline , 8 weeks
Change in cerebral oxygenation and perfusion as assessed by the Head-up tilt table testing (HUTT) with near-infrared spectroscopy (NIRS) monitoring. | Baseline , 8 weeks
Change in cognitive function as assessed by the NIH Toolbox assessment | Baseline , 8 weeks
  NIH Toolbox assessment evaluates multiple domains of cognitive performance including executive function, attention, episodic memory, language, processing speed, and working memory. Individual test scores are combined into a composite cognition score and reported as age-adjusted T-scores (mean = 50, SD = 10), where higher scores indicate better cognitive function.
Change in autonomic symptoms as assessed by the Composite Autonomic Symptom Score 31 (COMPASS-31) survey | Baseline , 8 weeks
  This is a 31 item questionnaire and each is scored from 0 (no symptoms) to 100(maximum symptom burden), with higher scores indicating more severe autonomic dysfunction.
Change in Impact of headaches as assessed by the Headache Impact Test (HIT-6) questionnaire | Baseline, 8 weeks
  HIT-6 questionnaire consists of 6 questions, each scored from 6(never) to 13(always), with total scores ranging from 36 to 78. Higher scores indicate a greater impact of headaches on quality of life.
Pulmonary function tests (PFTs), including spirometry and lung volume measurements | Baseline, 8 weeks
Change in Aortic diameter as assessed by the echocardiography | Baseline , 8 weeks

SECONDARY OUTCOMES:
Change in Levels of Nicotinamide adenine dinucleotide (NAD+) in whole blood as measured by high-performance liquid chromatography (HPLC) | Baseline , 8 weeks
Change in Levels of NR in whole blood as measured by high-performance liquid chromatography (HPLC) | Baseline , 8 weeks
Safety as assessed by number of participants that show drug toxicity as shown in bloodwork | Baseline
Safety as assessed by number of participants that show drug toxicity as shown in bloodwork | end of study (8 weeks after baseline)
Tolerability as assessed by the number of patients who complete study | end of study( 8 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Dianna Milewicz, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No